CLINICAL TRIAL: NCT06300138
Title: A Randomized Controlled Clinical Trial of Antifungal Agents and Infrared Thermotherapy Alone or in Combination in the Treatment of Sporotrichosis
Brief Title: Antifungal Agents and Infrared Thermotherapy Alone or in Combination in the Treatment of Sporotrichosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Gao Xinghua, Professor, First Hospital of China Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-631-2
Record Dates: First submitted 2024-02-29; First posted 2024-03-08 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-03

CONDITIONS: Sporotrichosis
Keywords: Sporotrichosis; local hyperthermia
MeSH Terms: conditions — Sporotrichosis | interventions — Itraconazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Drug combined with infrared hyperthermia group (Experimental): oral itraconazole (children less than 15 years old 6 mg/kg/d; adult patients: 200 mg/d) for a total course of 3-6 months, while infrared hyperthermia device for 3 consecutive days (times / day), each treatment for 30 minutes After two weeks (14 days), the lesions of the same target were treated continuously for 2 days (times per day), and then once a week for 2 consecutive times, the method was the same as before. After 7 times of treatment, the study physician decided whether to continue treatment n times after 1-2 weeks (n ≥ 0) according to the recovery of the subjects.
  Interventions: Other: Itraconazole and Infrared thermotherapy apparatus
- Drug group (Experimental): Itraconazole (6 mg/kg/d; for children less than 15 years old, 200 mg/d for adults) was taken orally for 3-6 months. The specific course of treatment was determined by the research physician according to the recovery of the subjects.
  Interventions: Drug: Itraconazole
- Infrared hyperthermia group (Experimental): Infrared hyperthermia device for 3 consecutive days (times / day), each treatment for 30 minutes After two weeks (14 days), the lesions of the same target were treated continuously for 2 days (times per day), and then once a week for 2 consecutive times, the method was the same as before. After 7 times of treatment, the study physician decided whether to continue treatment n times after 1-2 weeks (n ≥ 0) according to the recovery of the subjects.
  Interventions: Device: Infrared thermotherapy apparatus

INTERVENTIONS:
Drug: Itraconazole — oral itraconazole (children less than 15 years old 6 mg/kg/d; adult patients: 200 mg/d) for a total course of 3-6 months
  Arms: Drug group
Device: Infrared thermotherapy apparatus — infrared hyperthermia device for 3 consecutive days (times / day), each treatment for 30 minutes After two weeks (14 days), the lesions of the same target were treated continuously for 2 days (times per day), and then once a week for 2 consecutive times, the method was the same as before. After 7 times of treatment, the study physician decided whether to continue treatment n times after 1-2 weeks (n ≥ 0) according to the recovery of the subjects.
  Other Names: YY-WRY-V01 Infrared thermotherapy apparatus
  Arms: Infrared hyperthermia group
Other: Itraconazole and Infrared thermotherapy apparatus — oral itraconazole (children less than 15 years old 6 mg/kg/d; adult patients: 200 mg/d) for a total course of 3-6 months, while infrared hyperthermia device for 3 consecutive days (times / day), each treatment for 30 minutes After two weeks (14 days), the lesions of the same target were treated continuously for 2 days (times per day), and then once a week for 2 consecutive times, the method was the same as before. After 7 times of treatment, the study physician decided whether to continue treatment n times after 1-2 weeks (n ≥ 0) according to the recovery of the subjects.
  Arms: Drug combined with infrared hyperthermia group

SUMMARY:
Sporotrichosis is a chronic granulomatous mycosis caused by sporothrix complex. The course of sporotrichosis is always prolonged and even life-threatening, the treatment of this disease in an important scientific problem to be solved. The investigators previously found the predominance of subtype M2 macrophage which play an anti-inflammatory role in the lesions of sporotrichosis, the predominance of M2 macrophage may be responsible for the persistence of sporotrichosis; the investigators also found that local hyperthermia is effective in the treatment of sporotrichosis and hyperthermia treatment can activate the CRAC calcium channel in macrophages which triggers pro-inflammatory type M1 polarization and subsequent killing of sporothrix, however, the mechanism still calls for further investigation. The investigators hypothesize that hyperthermia leads to the activation of CRAC channels resulting in profound Ca2+ influx and Ca2+ upregulates NLRP3 inflammasome expression through inducing Nrf2 activation, then NLRP3 overexpression triggers M1 polarization and subsequent killing of sporothrix. Furthermore, the activation of Nrf2 upregulates STIM1 expression which forms a positive feedback for M1 type polarization of macrophages and further subsequent killing of sporothrix. The purpose of this project is to identify the hypothesis that hyperthermia could treat sporotrichosis by promoting pro-inflammatory type M1 polarization in macrophages, the mechanism by which hyperthermia could treat sporotrichosis is local hyperthermia could led to STIM1/CRAC calcium channel activation mediated calcium ions/Nrf2/NLRP3 induced M1 macrophages polarization and subsequent killing of sporothrix. The hypothesis will be identified at the cellular level, at the animal model level and at the clinical specimens level. The investigators believe that the project will guide the application of hyperthermia in the treatment of sporotrichosis and provide a new basis of theory and practice after the investigators achieving these goals.

ELIGIBILITY:
Inclusion Criteria:

* The results of pathology and fungal culture were all patients with sporotrichosis.
* Informed consent to the purpose and content of the study, and follow-up as required
* The physical condition and self-condition can cooperate with the treatment.

Exclusion Criteria:

* Subjects who are unable to maintain a relatively stable posture during treatment.
* Those who are sensitive or allergic to this experimental drug.
* Systemic antifungal or KI therapy within 12 months
* Local antifungal therapy within 1 month.
* Previous history of immunodeficiency virus (HIV) infection, or positive HIV antibody in screening period.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
the overall clinical clearance rate of skin lesions | Three months
  Three months after treatment, the overall clinical clearance rate of skin lesions in the three groups.

SECONDARY OUTCOMES:
Overall clinical clearance rate and recurrence rate | Six months
  Overall clinical clearance rate and recurrence rate of skin lesions in three groups
adverse reactions and incidence | Six months
  adverse reactions and incidence in three groups
the clearance rate of target skin lesions | Three months
  Three months after treatment, the clearance rate of target skin lesions in hyperthermia treatment group and hyperthermia combined with antifungal therapy group.
overall lesion clearance rate | Three months
  In patients with multiple lesions, the overall lesion clearance rate was 3 months after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of China Medical University, Shenyang, China

IPD SHARING:
Plan to Share IPD: No